CLINICAL TRIAL: NCT06105164
Title: Validation of a Novel Cerebellar-striatal Satiety Circuit in Humans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Mclean Hospital (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Laura M Holsen, Associate Professor of Psychiatry, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2023P002811
Record Dates: First submitted 2023-10-19; First posted 2023-10-27 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Appetitive Behavior; Obesity
MeSH Terms: conditions — Appetitive Behavior; Obesity | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active cerebellar rTMS (Active Comparator): Cerebellar targeted iTBS
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Sham cerebellar rTMS (Sham Comparator): Cerebellar targeted sham iTBS
  Interventions: Device: Sham repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — rTMS is a technique of TMS that allows for selective external manipulation of neural activity in a non-invasive manner. During rTMS a rapidly changing current is passed through an insulated coil placed against the scalp. This generates a temporary magnetic field, which in turn induces electrical current in neurons and allows for modulation of neural circuitry.
  Intermittent theta burst stimulation (iTBS) consisting of 2 s trains of 3 pulses at 50 Hz, repeated at 5 Hz, every 10s for a total of 600 pulses (82), will be applied to the target. Cerebellar stimulation will be applied to the targets at 100% of aMT or 35% maximal stimulator output, whichever is higher.
  Other Names: iTBS
  Arms: Active cerebellar rTMS
Device: Sham repetitive Transcranial Magnetic Stimulation (rTMS) — rTMS is a technique of TMS that allows for selective external manipulation of neural activity in a non-invasive manner. During rTMS a rapidly changing current is passed through an insulated coil placed against the scalp. This generates a temporary magnetic field, which in turn induces electrical current in neurons and allows for modulation of neural circuitry.
  Intermittent theta burst stimulation (iTBS) consisting of 2 s trains of 3 pulses at 50 Hz, repeated at 5 Hz, every 10s for a total of 600 pulses (82), will be applied to the target. Cerebellar stimulation will be applied to the targets at 100% of aMT or 35% maximal stimulator output, whichever is higher.
  Sham is achieved by using a coil with a magnetic shield preventing magnetic field from reaching the head.
  Other Names: iTBS
  Arms: Sham cerebellar rTMS

SUMMARY:
This study uses a noninvasive technique called transcranial magnetic stimulation (TMS) to study satiety in healthy individuals.

TMS is a noninvasive way of stimulating the brain, using a magnetic field to change activity in the brain. The magnetic field is produced by a coil that is held next to the scalp. In this study, the investigators will be stimulating the brain to learn more about the role of the cerebellum in satiety.

DETAILED DESCRIPTION:
The purpose of this study is to conduct a circuit manipulation experiment to test the hypothesis that targeting the cerebellum can alter activity in response to food cues to advance the understanding of the involvement of the cerebellar-striatal circuit in feeding behavior.

Participants will undergo an initial screening session to complete informed consent and undergo baseline assessments including physical activity and food craving. Participants will additionally undergo an MRI scan that includes structural and resting-state functional magnetic resonance imaging (rsfMRI). These rsfMRI imagines will be used to isolate individual resting state networks for targeting of rTMS modulation.

Participants will then complete two separate testing sessions involving MRI imaging and food intake assessments before and after rTMS. One visit will involve consumption of a filling meal; the other visit will be completed following an overnight fast.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged 18 to 65
* BMI of 20-35.0 kg/m2
* Normal or corrected-to-normal vision
* Good general health
* Ability to understand and willingness to sign written informed consent document

Exclusion Criteria:

* Current and/or past medical conditions
* Current and/or past eating disorder
* On a restricted diet and/or taking weight loss medication(s)
* History of bariatric surgery
* Weight fluctuation >3% in past 3 months
* Recent history of illicit recreational drug abuse
* Current nicotine use
* Intellectual disability
* Conditions that might result in increased risks of side effects or complications from TMS or MRI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Change in BOLD response in the cerebellum | 30 minutes pre-TMS and 30 minutes post-TMS, at each of two main study visits (fed, fasted)
  Change in functional activation of the cerebellum will be assessed before (pre-TMS) and after (post-rTMS) rTMS stimulation, measured separately at the fed visit and at the fasted visit.
Change in BOLD response in the ventral striatum | 30 minutes pre-TMS and 30 minutes post-TMS, at each of two main study visits (fed, fasted)
  Change in functional activation of the ventral striatum will be assessed before (pre-TMS) and after (post-rTMS) rTMS stimulation, measured separately at the fed visit and at the fasted visit.
Change in food reward valuation | up to 60 minutes pre-TMS and up to 60 minutes post-TMS, at each of two main study visits (fed, fasted)
  Change in food reward valuation of high-calorie foods will be assessed using the Willingness to Pay task, measured before (pre-TMS) and after (post-rTMS) rTMS stimulation, measured separately at the fed visit and at the fasted visit.
Ad libitum snack food intake | baseline, up to 60 minutes post-TMS at each of two main study visits (fed, fasted)
  Change in total caloric intake during the ad libitum snack food session will be assessed at the baseline visit and after (post-rTMS) rTMS stimulation, the latter measured separately at the fed visit and at the fasted visit.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Holsen, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - McLean Hospital, Belmont, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
Deidentified participant data will be shared with NIMH Data Repository (NDA).